CLINICAL TRIAL: NCT00115076
Title: A Phase IIIB Study to Evaluate the Mechanism of Action of 1.0 mg/kg Subcutaneously Administered Efalizumab in Adults With Moderate to Severe Plaque Psoriasis Who Are Candidates for Systemic Therapy
Brief Title: Study of the Drug Efalizumab (Raptiva), for Adult Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JKR-0511
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis
Keywords: skin; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — efalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- psoriasis (Experimental): moderate to severe plaque psoriasis
  Interventions: Drug: Efalizumab

INTERVENTIONS:
Drug: Efalizumab — 24 weekly doses of 1.0 mg/kg Efalizumab. Study drug will be administered by SC injection
  Other Names: Raptiva

SUMMARY:
Our laboratory is studying a skin disease known as psoriasis. The purpose of this protocol is to study the action and the effects of Efalizumab, on psoriasis. This medication has been studied extensively and has been found to be effective and safe in the treatment of psoriasis. The eligible patient will have 10% of his/her body surface area involved with psoriasis vulgaris.

DETAILED DESCRIPTION:
The eligible patient will receive the drug Efalizumab, weekly for 12 weeks, by injection. The patient will be seen weekly for 12 weeks and every other week for the 12 weeks of follow up. At those visits, the patient can expect that a physical and skin exam will be done. At specific weeks, blood work will be drawn, clinical photography taken and a skin biopsy done. Two types of skin biopsies will be done after local anesthesia has been administered. One is a punch biopsy where a small piece of skin will be taken, the approximate size of a pencil eraser. The second type of skin biopsy is shave biopsy, where a postage sized piece of skin will be taken.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent

* Plaque psoriasis covering >10% of total BSA
* Diagnosis of plaque psoriasis for at least 6 months
* PASI score >=12 (see Appendix A) or Linear PASI score of >= 8.0 at screening (see Appendix B)
* In the opinion of the investigator, candidate for systemic therapy for psoriasis:

  * Who has not been previously treated (naive to systemic treatment) OR
  * Who has had prior treatment with systemic therapy for psoriasis (e.g., PUVA, cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil (MMF), thioguanine, hydroxyurea, sirolimus, azathioprine, 6-MP, etanercept)
* Body weight of <140 kg
* 18 to 75 years old. As the risk of Efalizumab in childhood is unknown, those < 18years will be excluded from the study
* For women of childbearing potential or in men whose partners may become pregnant, willingness to use an acceptable method of contraception to prevent pregnancy for the duration of the study (while receiving study medication and 3 months following). Acceptable methods of contraception include use of a condom; abstinence; use by sexual partner of oral implantable or injectable contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap; or a sterile sexual partner
* Willingness to hold sun exposure reasonably constant and to avoid use of tanning booths or other UV light sources during the study

Exclusion Criteria

Subjects who meet any of the following exclusion criteria are ineligible for study entry:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* History of severe allergic or anaphylactic reactions to humanized monoclonal antibodies or fusion proteins that contain an Ig Fc region
* Clinically significant psoriasis flare during screening or on the first treatment day
* Treatment with efalizumab (anti-CD11a) within the last 12 months before enrollment
* Pregnancy or lactation. As the risk of Efalizumab in pregnancy is unknown, pregnant women will be excluded from the study
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of active tuberculosis (TB) or currently undergoing treatment for TB. PPD testing or chest X-ray is required for high-risk subjects (see Appendix D).

Subjects with a positive PPD (not due to BCG vaccination) or chest X-ray will be excluded

* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* Seropositivity for human immunodeficiency virus (HIV)
* Seropositivity for hepatitis B or C virus
* Hepatic enzymes >3 times the upper limits of normal (ULN)
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* WBC count <4000μL or >14,000/μL
* Serum creatinine >2 times the ULN
* Hospital admission for cardiac disease, stroke, or pulmonary disease within the last year
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders. Subjects with a history of fully resolved basal cell or squamous cell skin cancer may be enrolled
* History of substance abuse within the last 5 years
* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug Note: Certain medications and vaccines may not be used for specified periods of time prior to enrollment or at any time during the treatment period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-08-04 (Actual); Primary Completion 2009-05-18 (Actual); Study Completion 2011-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, Principal Investigator — Rockefeller University
Locations (2):
- United States (2):
  - Rockefeller University, New York, New York
  - The Rockefeller University, New York, New York

REFERENCES:
- [Derived] Johnson-Huang LM, Pensabene CA, Shah KR, Pierson KC, Kikuchi T, Lentini T, Gilleaudeau P, Sullivan-Whalen M, Cueto I, Khatcherian A, Hyder LA, Suarez-Farinas M, Krueger JG, Lowes MA. Post-therapeutic relapse of psoriasis after CD11a blockade is associated with T cells and inflammatory myeloid DCs. PLoS One. 2012;7(2):e30308. doi: 10.1371/journal.pone.0030308. Epub 2012 Feb 10. PMID 22348003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was not assigned to any arm.
Period: Overall Study
Arm/Group | Psoriasis
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: years
Arm/Group | Psoriasis
Number analyzed (Participants) | 30
Number analyzed (years) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Improvement of Target Lesions
Description: a single composite score based on quantitative measurement of epidermal acanthosis, qualitative expression of Keratin16 (histochemistry assessment) and quantitative measurement of K16 mRNA.
Time Frame: week 12
Population: 28 out of 30 participants completed the study. Then clinical improvement was determined only for those 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Psoriasis
Number analyzed (Participants) | 28
Participants | 18

2. Secondary Outcome: Assessment of Overall Clinical Response as Measured by Psoriasis Area and Severity Index (PASI)
Description: Psoriasis Area and Severity Index (PASI) combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). Clinical response defined as PASI improvement over 75% at week 12.
Time Frame: Day 0, day 14, day 42, day 84, Days 112, 140, and 168. PASI has been measured at those timepoints but outcome is related to Baseline and Day 84.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriasis
Number analyzed (Participants) | 30
score on a scale
  Baseline | 34.58 (17.48)
  Week 12 | 12.94 (10.68)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Psoriasis
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 9/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psoriasis (N=30)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 9 (9)
fatigue (General disorders) | 9 (9)
diarrhea (Gastrointestinal disorders) | 4 (4)
joint pain (Musculoskeletal and connective tissue disorders) | 6 (6)
dizziness (General disorders) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
dry mouth (Gastrointestinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
aphthous ulcer (Gastrointestinal disorders) | 1 (1)
chills (General disorders) | 4 (4)
headache (General disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 2 (2)
fever (General disorders) | 4 (4)
abdominal pain (Gastrointestinal disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes